CLINICAL TRIAL: NCT02096549
Title: Validity of Bispectral Index Monitoring During Deep Sedation for Botulinum Toxin Injection in Children With Cerebral Palsy
Brief Title: Validity of Bispectral Index Monitoring During Deep Sedation
Status: Completed | Type: Observational
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Sung Mee Jung, Associate professor in Anesthesiology and Pain Medicine, Yeungnam University College of Medicine
Other Study IDs: YUH-14-0319-O10
Record Dates: First submitted 2014-03-17; First posted 2014-03-26 (Estimated); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; Botulinum toxin; Propofol; Deep sedation; Bispectral index monitor
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During Intramuscular botulinum toxin injections for children with cerebral palsy, immobility is essential to inject botulinum toxin to the right muscle. Because children with cerebral palsy are generally unable to control their movement, deep sedation is required during this painful procedure.

Short-acting drugs such as propofol and remifentanil are widely used for pediatric anesthesia and sedation but still have possibility of over-sedation and associated complications due to their rather narrow therapeutic window. Therefore, objective scoring system to assess the level of sedation to provide an effective and safe sedation in children. Bispectral index (BIS) monitoring,an objective guidance of sedation might be helpful.

The present study is to investigate the validity of the BIS monitoring during deep sedation of children with cerebral palsy for injection of botulinum toxin.

DETAILED DESCRIPTION:
Intramuscular botulinum toxin injections for children with cerebral palsy have been extensively performed to relive spasticity and improve rehabilitation. During procedure immobility is essential to inject botulinum toxin to the right muscle for optimal effect. Because children with cerebral palsy are generally unable to control their movement, deep sedation is required during this painful procedure.

Short-acting drugs with rapid, predictable onset and offset of action, such as propofol and remifentanil, facilitate infusion rate adjustments and rapid recovery. However, there is always the possibility of over-sedation, hypotension and respiratory depression due to their rather narrow therapeutic window.

Several clinical sedation scales have been used to provide an effective and safe sedation in children. Because clinical scoring depends on patient response to verbal or physical stimulation, it is difficult to assess the level of sedatin in patients with deep sedation during delicate phase of the procedure. Bispectral index (BIS) monitoring,an objective guidance of sedation might be helpful. Although BIS scores in children with conscious and deep sedation were reported to correlate with clinical sedation scales, the validity during painful procedure in children with cerebral palsy was not investigated yet.

The present study is to investigate the validity of the BIS monitoring and its correlation to University of Michigan sedation scale during deep sedation of children with cerebral palsy for injection of botulinum toxin.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-II healthy children Ages Eligible for study: 3 to 18 years scheduled for injection of botulinum toxin under deep sedation

Exclusion Criteria:

* Unstable cardiac disease Recent (< 8 week) pneumonia, bronchitis, asthma attack, respiratory infection Craniofacial defect History of a difficult airway management Hypotonia and lack of head control Tremors

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: primary care clinic (rehabilitation)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duk Hee Lee, M.D., Study Director — Yeungnam University Hospital
Locations (1):
- Yeungnam University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No
no plan to share our data

REFERENCES:
- [Background] McDermott NB, VanSickle T, Motas D, Friesen RH. Validation of the bispectral index monitor during conscious and deep sedation in children. Anesth Analg. 2003 Jul;97(1):39-43, table of contents. doi: 10.1213/01.ane.0000067402.02136.a2. PMID 12818940
- [Background] Soudant DL, Staal HM, Witlox AM, Vles JS. Conscious sedation or general anaesthetic for intramuscular botulinum toxin injections in children - a two centre cross-sectional prospective audit. Eur J Paediatr Neurol. 2013 Mar;17(2):219-20. doi: 10.1016/j.ejpn.2012.06.012. Epub 2012 Aug 4. No abstract available. PMID 22871256
- [Background] American Academy of Pediatrics; American Academy of Pediatric Dentistry; Cote CJ, Wilson S; Work Group on Sedation. Guidelines for monitoring and management of pediatric patients during and after sedation for diagnostic and therapeutic procedures: an update. Paediatr Anaesth. 2008 Jan;18(1):9-10. doi: 10.1111/j.1460-9592.2007.02404.x. No abstract available. PMID 18095958

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at Yeungnam Univerisity Hospital in South korea from March 2014 to April 2017. Twenty children with spastic CP, with an American Society of Anesthesiologists physical status of 1 and 2, aged between 3 and 18 years, who were scheduled for a botulinum toxin injection under deep sedation, were enrolled.
Pre-assignment Details: This prospective observational study was approved by the Institutional Review Board (YUH-14-0319-O10) and was registered with ClinicalTrials.gov (NCT02096549) on March 28, 2014. Written informed consent from the participants' parents and, when appropriate, verbal assent from the participating children were obtained before enrollment in the study.
Groups:
- Children With Spastic Cerebral Palsy: children with spastic CP, with an American Society of Anesthesiologists physical status of 1 and 2, aged between 3 and 18 years, who were scheduled for a botulinum toxin injection under deep sedation, were enrolled. Children were excluded from the study if they had an anticipated difficult airway, unstable cardiac disease, craniofacial defect, allergy to drugs used in this study, and/or history of recent (< 8 weeks) pneumonia, bronchitis, asthma attack, or an upper respiratory infection.
Period: Overall Study
Arm/Group | Children With Spastic Cerebral Palsy
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 22 children with cerebral palsy
Groups:
- Spastic Cerebral Palsy: After confirmation of adequate spontaneous respiration 5 minutes after remifentanil infusion in children, an attending anesthesiologist administered propofol (1.5 mg/kg) mixed with lidocaine (1 mg/kg) over 1 minute followed by continuous infusion of propofol on the basis of clinical signs of arousability, movement, blood pressure, heart rate and respiratory rate. Two independent investigators, who were blinded to BIS values, assessed the level of sedation using the UMSS scores every minute from baseline to induction of deep sedation. BIS values measured immediately before stimulation for assessing the UMSS observation were collected by another independent investigator. The BIS value with a signal quality index (SQI) ≥ 50 was accepted for analysis. Spearman rank order correlation analysis was used to evaluate the relationship of BIS and UMSS. The cut-off BIS value for detecting deep sedation was determined by analysis of receiver-operating characteristic (ROC) curve. The area under the
Arm/Group | Spastic Cerebral Palsy
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.5 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  sex: Female | 7
  sex: Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 20

OUTCOME MEASURES:

1. Primary Outcome: The Correlation Between the Paired BIS Value Categories and Clinical Sedation Scores
Description: Two independent investigators assessed the level of sedation using the Universtiy of Michigan sedation scale (UMSS) and modified observer's assessment of alertness and sedation (MOAAS) scales every 1 min during the induction of sedation and every 3 min during the maintenance of sedation. The BIS values at each UMSS and MOAAS score were collected. The correlation between the BIS score and UMSS score, and BIS score and MOAAS score was analyzed using the Spearman rank correlation test. The correlation coefficient is expressed as an r-value, and this value is expressed as a single value, not as a range with the lowest and highest values. The higher the value, the better the outcome.
Time Frame: From induction of sedation to completion of procedure(botulinum toxin injection)
Population: Children with spastic Cerebral Palsy undergoing botulinum toxin injection
Measure: Number (97.5% Confidence Interval); unit: correlation coefficient
Arm/Group | Children With Spastic Cerebral Palsy
Number analyzed (Participants) | 20
correlation coefficient
  correlation of the UMSS score and BIS value | 0.917 [0.858 to 0.969]
  Correlation for the MOAAS score and BIS value | 0.874 [0.808 to 0.940]

ADVERSE EVENTS:
Time Frame: 24 hours
Groups:
- Validity of Bispectral Index Monitoring: After confirmation of adequate spontaneous respiration 5 minutes after remifentanil infusion in children, an attending anesthesiologist administered propofol (1.5 mg/kg) mixed with lidocaine (1 mg/kg) over 1 minute followed by continuous infusion of propofol on the basis of clinical signs of arousability, movement, blood pressure, heart rate and respiratory rate. Two independent investigators, who were blinded to BIS values, assessed the level of sedation using the UMSS scores every minute from baseline to induction of deep sedation. BIS values measured immediately before stimulation for assessing the UMSS observation were collected by another independent investigator. The BIS value with a signal quality index (SQI) ≥ 50 was accepted for analysis. Spearman rank order correlation analysis was used to evaluate the relationship of BIS and UMSS. The cut-off BIS value for detecting deep sedation was determined by analysis of receiver-operating characteristic (ROC) curve. The area under the
Arm/Group | Validity of Bispectral Index Monitoring
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
This study has some limitations. We couldn't identify the age-related correlations among the CP children undergoing botulinum toxin injection and we did not know the correlation with BIS scores and UMSS and MOAAS scores according to sex.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-30): https://cdn.clinicaltrials.gov/large-docs/49/NCT02096549/Prot_SAP_000.pdf